CLINICAL TRIAL: NCT00409578
Title: A Randomized, Double-blind, Parallel-group, Placebo-controlled, Multinational Clinical Trial to Evaluate the Efficacy of Aliskiren and Valsartan Versus Placebo in Lowering Levels on NT-proBNP in Stabilized Patients Post Acute Coronary Syndromes
Brief Title: Efficacy and Safety of Aliskiren and Valsartan Versus Placebo in Patients Stabilized Following an Acute Coronary Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: The TIMI Study Group (Other)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSPP100A2347
Record Dates: First submitted 2006-12-07; First posted 2006-12-11 (Estimated); Results first posted 2011-02-02 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Post Acute Coronary Syndrome; Myocardial Ischemia
Keywords: Post acute coronary syndrome; Acute; coronary syndrome; B-type natriuretic peptide; N-terminal; pro-B-type natriuretic peptide; myocardial infarctions
MeSH Terms: conditions — Myocardial Ischemia; Angina, Unstable; Myocardial Infarction | interventions — aliskiren; Valsartan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- Placebo (Placebo Comparator): Placebo tablets and capsules
  Interventions: Drug: Placebo
- Aliskiren 300 mg (Experimental): Following 1 week of treatment with 75 mg of aliskiren (tablets), patients in this arm were titrated up to 150 mg of aliskiren; 1 week later they were titrated up to 300 mg aliskiren for the remainder of the study.
  Interventions: Drug: Aliskiren 300 mg
- Valsartan 320 mg (Experimental): Following 1 week of treatment with 80 mg of valsartan (capsules), patients in this arm were titrated up to 160 mg of valsartan; 1 week later they were titrated up to 320 mg valsartan for the remainder of the study.
  Interventions: Drug: Valsartan 320 mg
- Aliskiren/valsartan 300/320 mg (Experimental): Following 1 week of treatment with 80 mg of valsartan (capsules), patients in this arm were titrated up to 160 mg of valsartan; 1 week later they were titrated up to 320 mg valsartan for the remainder of the study. Beginning with Week 4, in addition to 320 mg valsartan, patients were treated with 75 mg of aliskiren (tablets); 1 week later patients were titrated up to 150 mg of aliskiren and 1 week later they were titrated up to 300 mg aliskiren for the remainder of the study.
  Interventions: Drug: Aliskiren/valsartan 300/320 mg

INTERVENTIONS:
Drug: Placebo — Placebo tablets and capsules. In order to adequately blind the study, patients were required to take a total of 1 tablet and 2 capsules during the first 4 weeks of the study. During the remainder of the study, patients were required to take 2 tablets and 2 capsules. Each dose was taken by mouth with water at approximately 8:00 AM with or without food.
  Arms: Placebo
Drug: Aliskiren 300 mg — Following 1 week of treatment with 75 mg of aliskiren (tablets), patients in this arm were titrated up to 150 mg of aliskiren; 1 week later they were titrated up to 300 mg aliskiren for the remainder of the study. If a patient was not up-titrated or required down-titration, the patient continued on that dose for the remainder of the study. If 2 down-titrations were required, they stopped study drug. In order to adequately blind the study, patients were required to take 1 tablet and 2 capsules during the first 4 weeks of the study and 2 tablets and 2 capsules for the remainder of the study. Each dose was taken by mouth with water at approximately 8:00 AM.
  Arms: Aliskiren 300 mg
Drug: Valsartan 320 mg — Following 1 week of treatment with 80 mg of valsartan (capsules), patients in this arm were titrated up to 160 mg of valsartan; 1 week later they were titrated up to 320 mg valsartan for the remainder of the study. If a patient was not up-titrated or required down-titration, the patient continued on that dose for the remainder of the study. If 2 down-titrations were required, they stopped study drug. In order to adequately blind the study, patients were required to take 1 tablet and 2 capsules during the first 4 weeks of the study and 2 tablets and 2 capsules for the remainder of the study. Each dose was taken by mouth with water at approximately 8:00 AM.
  Arms: Valsartan 320 mg
Drug: Aliskiren/valsartan 300/320 mg — Following 1 week of treatment with 80 mg of valsartan (capsules), patients in this arm were titrated up to 160 mg of valsartan; 1 week later they were titrated up to 320 mg valsartan for the remainder of the study. Beginning with Week 4, in addition to 320 mg valsartan, patients were treated with 75 mg of aliskiren (tablets); 1 week later patients were titrated up to 150 mg of aliskiren and 1 week later they were titrated up to 300 mg aliskiren for the remainder of the study. If a patient was not up-titrated or required down-titration, the patient continued on that dose for the remainder of the study. If 2 down-titrations were required, they stopped study drug. In order to adequately blind the study, patients were required to take 1 tablet and 2 capsules during the first 4 weeks of the study and 2 tablets and 2 capsules for the remainder of the study. Each dose was taken by mouth with water at approximately 8:00 AM.
  Arms: Aliskiren/valsartan 300/320 mg

SUMMARY:
The purpose of this study is to test the hypothesis that the inhibition of the renin-angiotensin-aldosterone system (RAAS) with the angiotensin receptor blocker valsartan or the renin antagonist aliskiren will improve ventricular hemodynamics, as reflected by a greater reduction in levels of N-terminal proB-type natriuretic peptide (NT-proBNP) compared to placebo in subjects stabilized following acute coronary syndrome (ACS) who are determined to be at high risk due to an elevated concentration of natriuretic peptides.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients 18 years old or older
* Subjects who are hospitalized for ischemic chest discomfort at rest lasting at least 10 minutes and consistent with cardiac ischemia
* Final diagnosis of acute coronary syndrome
* Elevated concentrations of natriuretic peptide 3-10 days after admission for their qualifying acute coronary syndrome event

Exclusion Criteria:

* Known or suspected contraindications, including history of allergy or hypersensitivity to angiotensin receptor blockers (ARBs), renin antagonists, or to drugs with similar chemical structures.
* Presence of clinically overt heart failure
* Known evidence of left ventricular systolic dysfunction
* Percutaneous coronary intervention (PCI) less than 24 hours before randomization.
* Patients on chronic ACEI or ARB therapy for whom therapy with an ACEI or ARB is clinically required with no reasonable alternative therapy available.

Other protocol-defined inclusion/exclusion criteria applied to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1101 (Actual)
Dates: Start 2007-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Braunwald, MD, Study Chair — TIMI Study Group, Boston, MA
Locations (11):
- Investigative Site, Investigative Site, New Jersey, United States
- Investigative Site, Investigative Site, Belgium
- Investigative Site, Investigative Site, Canada
- Investigative Site, Investigative Site, Czechia
- Investigative Site, Investigative Site, Germany
- Investigative Site, Investigative Site, Hungary
- Investigative Site, Investigative Site, Netherlands
- Investigative Site, Investigative Site, Poland
- Investigative Site, Investigative Site, Russia
- Investigative Site, Investigative Site, Spain
- Investigative Site, Investigative Site, Sweden

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Aliskiren 300 mg | Valsartan 320 mg | Aliskiren/Valsartan 300/320 mg
Started | 280 | 271 | 269 | 281
Completed | 228 | 201 | 215 | 214
Not Completed | 52 | 70 | 54 | 67
Not completed — Adverse Event | 27 | 37 | 25 | 33
Not completed — Abnormal laboratory value(s) | 2 | 2 | 2 | 4
Not completed — Lack of Efficacy | 0 | 0 | 0 | 2
Not completed — Subject no longer requires study drug | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 8 | 15 | 16 | 17
Not completed — Lost to Follow-up | 2 | 0 | 2 | 2
Not completed — Administrative problems | 8 | 9 | 2 | 4
Not completed — Death | 2 | 4 | 4 | 2
Not completed — Protocol Violation | 3 | 2 | 3 | 1
Not completed — Missing | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Aliskiren 300 mg | Valsartan 320 mg | Aliskiren/Valsartan 300/320 mg | Total
Number analyzed (Participants) | 280 | 271 | 269 | 281 | 1101
Age Continuous [Mean (Standard Deviation); unit: years] | 63 (11.8) | 63 (11.7) | 64 (11.6) | 63 (11.1) | 63 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 86 | 72 | 87 | 348
  Male | 177 | 185 | 197 | 194 | 753

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in N-terminal proB-type Natriuretic Peptide (NT-proBNP) at Week 8
Description: Blood samples for the measurement of NT-proBNP were collected, processed, and shipped to the TIMI Biomarker Core Laboratory, Boston MA for storage and analysis. The change from baseline to Week 8 was expressed as the geometric mean of the ratio: Week 8/Baseline.
Time Frame: Baseline to Week 8
Population: Full analysis set: All patients who were correctly randomized. Missing baseline values were not imputed. The last post-baseline biomarker measurement collected was used for analysis. In the aliskiren treated group, 4 patients never received study drug but were included in the full analysis set but were not included in any efficacy analyses.
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Placebo | Aliskiren 300 mg | Valsartan 320 mg | Aliskiren/Valsartan 300/320 mg
Number analyzed (Participants) | 259 | 235 | 246 | 256
pg/mL | 0.582 [0.502 to 0.676] | 0.563 [0.483 to 0.656] | 0.614 [0.526 to 0.716] | 0.635 [0.548 to 0.737]

2. Secondary Outcome: Change From Baseline in B-type Natriuretic Peptide (BNP) at Week 8
Description: Blood samples for the measurement of BNP were collected, processed, and shipped to the TIMI Biomarker Core Laboratory, Boston MA for storage and analysis. The change from baseline to Week 8 was expressed as the geometric mean of the ratio: Week 8/Baseline.
Time Frame: Baseline to Week 8
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Placebo | Aliskiren 300 mg | Valsartan 320 mg | Aliskiren/Valsartan 300/320 mg
Number analyzed (Participants) | 252 | 229 | 237 | 252
pg/mL | 0.642 [0.535 to 0.770] | 0.597 [0.495 to 0.720] | 0.670 [0.554 to 0.810] | 0.682 [0.568 to 0.818]

3. Secondary Outcome: Percentage of Patients With a Cardiac Event
Description: A cardiac event was defined as at least one of the following events: Cardiovascular death, recurrent myocardial infarction (MI), or hospitalization for congestive heart failure (CHF), all to be confirmed by adjudication.
Time Frame: Baseline to Week 8
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Placebo | Aliskiren 300 mg | Valsartan 320 mg | Aliskiren/Valsartan 300/320 mg
Number analyzed (Participants) | 278 | 268 | 268 | 278
Percentage of patients | 2.9 | 4.9 | 4.9 | 4.0

4. Secondary Outcome: Percentage of Patients With a Composite Clinical-biochemical Event
Description: A composite clinical-biochemical event was defined as at least one of the following events: cardiovascular death confirmed by adjudication, recurrent MI confirmed by adjudication, hospitalization for CHF confirmed by adjudication, and/or NT-proBNP => 200 pg/mL.
Time Frame: Baseline to Week 8
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Placebo | Aliskiren 300 mg | Valsartan 320 mg | Aliskiren/Valsartan 300/320 mg
Number analyzed (Participants) | 278 | 268 | 268 | 278
Percentage of patients | 79.5 | 73.5 | 77.2 | 75.2

ADVERSE EVENTS:
Description: Safety set: All patients that received at least 1 dose of study drug. Missing values were not imputed. In the aliskiren group, 4 patients were excluded because they never received study drug. One patient who never received study drug was included in the safety set because he had a date for the end of study treatment on the study completion page.
Arm/Group | Placebo | Aliskiren 300 mg | Valsartan 320 mg | Aliskiren/Valsartan 300/320 mg
Serious Adverse Events (participants affected / at risk) | 26/278 | 39/264 | 33/268 | 46/279
Other Adverse Events (participants affected / at risk) | 64/278 | 61/264 | 51/268 | 57/279
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=278) | Aliskiren 300 mg (N=264) | Valsartan 320 mg (N=268) | Aliskiren/Valsartan 300/320 mg (N=279)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 3 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 4 | 2 | 0
Angina pectoris (Cardiac disorders) | 2 | 5 | 3 | 6
Angina unstable (Cardiac disorders) | 1 | 2 | 1 | 4
Atrial fibrillation (Cardiac disorders) | 2 | 1 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 2 | 1 | 3 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 2 | 2 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 1
Dressler's syndrome (Cardiac disorders) | 1 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 2 | 0 | 5
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 1 | 4
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 1 | 0
Postinfarction angina (Cardiac disorders) | 1 | 0 | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0
Cardiac death (General disorders) | 0 | 0 | 1 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 7 | 2 | 3
Sudden cardiac death (General disorders) | 0 | 2 | 2 | 0
Sudden death (General disorders) | 1 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 2 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1
Helicobacter gastritis (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 3 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0
Arterial injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Thrombosis in device (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
ECG signs of myocardial ischaemia (Investigations) | 1 | 0 | 0 | 0
Heart rate decreased (Investigations) | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypoglycaemic unconsciousness (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 2
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1 | 0
Arterial occlusive disease (Vascular disorders) | 0 | 1 | 0 | 0
Arterial stenosis (Vascular disorders) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Femoral artery aneurysm (Vascular disorders) | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Hypertensive emergency (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 3 | 0 | 2
Ischaemia (Vascular disorders) | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=278) | Aliskiren 300 mg (N=264) | Valsartan 320 mg (N=268) | Aliskiren/Valsartan 300/320 mg (N=279)
Angina pectoris (Cardiac disorders) | 13 | 9 | 14 | 8
Hyperkalaemia (Metabolism and nutrition disorders) | 17 | 16 | 13 | 13
Dizziness (Nervous system disorders) | 15 | 23 | 13 | 19
Headache (Nervous system disorders) | 18 | 10 | 7 | 10
Orthostatic hypotension (Vascular disorders) | 14 | 16 | 12 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.